CLINICAL TRIAL: NCT04346849
Title: Tooth Discoloration Induced by Different Calcium Silicate Based Materials: in Vivo Study
Brief Title: Tooth Discoloration Induced by Pulpotomy Materials
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Nessrin Taha, Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5/2018
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Tooth Discoloration
Keywords: Pulpotomy, MTA, Biodentine, Bioceramic, discoloration
MeSH Terms: conditions — Tooth Discoloration | interventions — Pulpotomy

STUDY DESIGN:
Intervention Model Description: Three groups will receive the same treatment procedure but randomly assigned to one of three different materials, tooth color changes will be measured at certain time points and will be compared between the 3 groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant will not be informed about the type of material. Investigator will be given the material only after the pulpotomy procedure was completed according to a random sequence number generator. Upon tooth color measurement the investigator will not be informed about the type of material
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MTA pulpotomy (Experimental): Teeth receiving pulpotomy using MTA
  Interventions: Procedure: Pulpotomy
- Biodentine pulpotomy (Experimental): Teeth receiving pulpotomy using Biodentine
  Interventions: Procedure: Pulpotomy
- Bioceramic pulpotomy (Experimental): Teeth receiving pulpotomy using Bioceramic
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: Pulpotomy — Cutting the coronal portion of the pulp and application of a calcium silicate based material followed by restoration

SUMMARY:
Vital pulp therapy including pulpotomy is commonly used for managing teeth with carious pulp exposure instead of performing root canal therapy. The gold standard materials used in this procedure are the calcium silicate based materials, however recent case reports have shown tooth discoloration caused by these materials especially MTA which is of concern to the patients. The aim of this study is to compare tooth color changes and discoloration induced by 3 calcium silicate based materials used in pulpotomy over 6 months, 12 months and yearly up to 5 years.

DETAILED DESCRIPTION:
Pulpotomy procedure involves removal of the coronal portion of the dental pulp followed by placement of a compatible material and subsequent coronal restoration of the tooth. Mineral trioxide aggregate is the gold standard material used in pulpotomy; however it has been implicated in tooth discoloration due to it radioopacifier. newer calcium silicate based materials including Biodentine and bioceramic have different opacifier and claimed not to cause tooth discoloration in laboratory studies.

In this clinical study tooth color measurement of teeth treated by pulpotomy using these 3 materials will be taken using vita easy shade device immediately after placement of the materials, 6 months and 12 months after the treatment then yearly up to 5 years. The discoloration potential of these 3 materials will be compared. Factors that may influence tooth discoloration will be also measured and analyzed including buccal wall thickness and time of bleeding control after pulpotomy.

ELIGIBILITY:
Inclusion Criteria:

* Vital tooth with carious pulp exposure to be treated by full pulpotomy
* Fully erupted upper or lower molar tooth with fully formed apex
* Tooth should have intact buccal wall (no caries or restoration)
* Tooth should be restorable by direct composite restoration

Exclusion Criteria:

* Partially erupted tooth
* Tooth has caries on the buccal surface
* Tooth has restoration on buccal surface
* Tooth has preoperative coronal staining compared to adjacent teeth

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-09-02 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
Tooth color change | Immediate, 6 months, 1 year and yearly up to 5 years
  Darkening in tooth color shade after placement of the calcium silicate based material

CONTACTS AND LOCATIONS:
Overall Officials: Nessrin Taha, DCD, Study Chair — Jordan University of Science and Technology
Locations (2):
- Jordan (2):
  - Dental teaching centre Faculty Of Dentistry, Irbid
  - Jordan University of science and technology, Irbid

IPD SHARING:
Plan to Share IPD: No
The data will be shared in the publication of the 1 year results of the study. If furthers details or data required the study chair can be contacted by email

REFERENCES:
- [Derived] Taha NA, Hamdan AM, Al-Hiyasat AS. Coronal discoloration induced by calcium silicate-based cements used in full pulpotomy in mature permanent molars: a randomized clinical trial. Clin Oral Investig. 2023 Apr;27(4):1723-1730. doi: 10.1007/s00784-022-04799-x. Epub 2022 Nov 29. PMID 36445467